CLINICAL TRIAL: NCT00629772
Title: A Double-Blind Study on the Safety and Efficacy of Infliximab in Palmoplantar Psoriasis
Brief Title: Safety and Efficacy of Infliximab in Palmoplantar Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inno-6003; P-05121 (Other: Schering Plough Canada)
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Results first posted 2010-09-02 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Palmoplantar Psoriasis
Keywords: Palmoplantar psoriasis; Infliximab
MeSH Terms: interventions — Sodium Chloride; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo then infliximab (Placebo Comparator): Placebo at weeks 0, 2, 6 during the first intervention period and infliximab 5mg/kg at weeks 14, 16 and 20 during second intervention period.
  Interventions: Drug: Placebo; Drug: Infliximab
- Infliximab (Active Comparator): Infliximab 5mg/kg at weeks 0, 2, 6, 14 and 22.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Placebo — Patients receive placebo on weeks 0, 2 and 6. They receive infliximab 5mg/kg at weeks 14, 16 and 20.
  Other Names: Saline
  Arms: Placebo then infliximab
Drug: Infliximab — Patients in infliximab group receive infliximab 5mg/kg at weeks 0, 2, 6, 14 and 22. Patients in placebo then infliximab group receive placebo at weeks 0, 2, 6, then receive infliximab at weeks 14, 16 and 20.
  Other Names: Remicade

SUMMARY:
Palmoplantar psoriasis is a variant of psoriasis affecting palms and soles. It is one of the most debilitating variants of psoriasis which very often interferes with daily activities and with the ability to work. This type of psoriasis is very difficult to treat as topicals have difficulty penetrating the thick epidermis of palms and soles and are therefore not very effective. The response to standard agents (methotrexate, cyclosporine and acitretin) is also usually limited. A number of these patients have very severe hand and feet disease with mild to no involvement elsewhere on the body.

Given the efficacy of infliximab in psoriasis, the purpose of this study is to evaluate if infliximab is safe and if it will improve severity and quality of life in patients with palmoplantar psoriasis, a debilitating variant of psoriasis.

DETAILED DESCRIPTION:
A total of 24 patients with non-pustular palmoplantar psoriasis affecting at least 10% of the combined palms and soles area and with a modified palmoplantar pustulosis area severity index (m-PPPASI) of at least 8 will be recruited. Patients will be randomized (1:1) to receive either infliximab 5 mg/kg or placebo (normal saline) on weeks 0, 2 and 6. Patients assigned to placebo during the first 3 infusions will receive infliximab 5 mg/kg at weeks 14, 16 and 20 and placebo again at week 22 while patients who were assigned to receive infliximab during the first 3 infusions will receive infliximab at week 14 and placebo at week 16 and week 20 as well as infliximab for the last infusion at week 22. The primary endpoint will be at week 14. Patients will come back to the clinic at week 26 for a final efficacy and safety assessment.

Efficacy will be evaluated by assessing psoriasis plaque severity on palms and soles (physician's global assessment PGA), percentage of palms and soles area affected by psoriasis (palmoplantar surface area - PPSA) as well as m-PPPASI (modified palmoplantar pustulosis area and severity index). Quality of life will be evaluated at every visit by performing the dermatology life quality index DLQI. Safety will be evaluated by repeating chemistry and haematology laboratories at regular visits as well as by physical examinations and assessment of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient has a history of palmoplantar psoriasis for at least 6 months.
* Patient has a m-PPPASI of at least 8 with at least 10% of the total surface of palms and soles affected with psoriasis at baseline
* Patients who failed either 4 weeks (or more) of treatment with a potent or superpotent topical corticosteroid, methotrexate, acitretin, cyclosporine, efalizumab, etanercept or alefacept for the treatment of palmoplantar psoriasis. Patients with a positive PPD who accept TB prophylaxis, will need to have failed 4 weeks (or more) of treatment with methotrexate, acitretin, cyclosporine, efalizumab, etanercept, alefacept or any other systemic therapies for the treatment of palmoplantar psoriasis.
* Patient with a history and/or the presence of typical plaque psoriasis outside palms and soles
* Female patient is either not of childbearing potential or is of childbearing potential and practicing an acceptable contraception
* Female patients of childbearing potential must have a negative serum pregnancy test at the Screening visit.
* Patient is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, and physical examination performed at Screening
* The investigator evaluates that the benefit / risk ratio is acceptable for the patient.
* Patients must be able and willing to provide written informed consent and comply with the requirements of this study protocol.
* Negative PPD
* Patients with a positive PPD may be eligible if they initiate TB prophylaxis before the first injection of infliximab

Exclusion Criteria:

* Patient has a history of pustules on palms and/or soles or currently has evidence of pustules on palms and/or soles.
* Patient with Chest X Ray findings positive or suspicious for active tuberculosis.
* Patient has had opportunistic infections.
* Patient has had active TB or recent close contact with an individual with active TB.
* Patient has had a serious infection, has been hospitalized for an infection, or has been treated with intravenous (IV) antibiotics for an infection within 2 months prior to Day 0.
* Patient has had a chronic or recurrent infectious disease including hepatitis B or hepatitis C.
* Patient has a known malignancy or history of malignancy within 5-year period prior to screening (with the exception of squamous or basal cell carcinoma of the skin that has been completely excised without evidence of recurrence).
* Patient has a history of lymphoproliferative disease, has multiple sclerosis, or other central demyelinating disorder, or congestive heart failure.
* Patient has elevated aspartate aminotransferase or alanine aminotransferase levels more than twice the upper limit of normal at screening.
* Patient has received live vaccination within 3 months of randomization or plans to receive live vaccination during the study or within 3 months after the last infusion.
* Patient is pregnant, breastfeeding, or planning pregnancy (both men and women) during the trial or within the 6-month period thereafter.
* Patient has a history of an allergic reaction to infliximab or any constituent of study drug.
* Patient who has used any topical treatment for psoriasis (except non-medicated emollients) in the last 2 weeks before Day 0 with the exception of hydrocortisone and desonide for the face, groin (including genitals) and inframammary areas as well as shampoos containing tar, salicylic acid or zinc pyrithione
* Patient who has used UVB phototherapy or excessive sun exposure less than 14 days before Day 0.
* Patient has used any non-biological systemic therapy for the treatment of psoriasis (including PUVA therapy), systemic steroids or systemic immunosuppressants less than 28 days before Day 0. Investigational non-biologics agents must be discontinued at least 28 days or 5 half-lives prior to Day 0 (whichever is longer).
* Patient is currently participating in a clinical trial with an experimental drug or device.
* Patient who has used any biological therapy for the treatment of psoriasis less than 90 days before day 0.
* Patient is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed. Patients who have used oral or injectable corticosteroids less than 28 days before Day 0 are excluded.
* Patient has a poorly controlled medical condition which, in the opinion of the investigator, would put the patient at risk if the patient participated in the study.
* Patient currently uses or plans to use anti-retroviral therapy at any time during the study.
* Patient is known to have immune deficiency or is immunocompromised.
* Patient is known to be infected with the human immunodeficiency virus, hepatitis B or hepatitis C virus.
* Patient has current signs or symptoms or has a history of systemic lupus erythematosus.
* Patient has a history of clinically significant drug or alcohol abuse in the last year.
* Patient has erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis.
* Patients with a positive PPD who accept TB prophylaxis must not have any pre-existing liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research
Locations (5):
- Canada (5):
  - The Guenther Dermatology Research Center, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - Innovaderm Research Laval, Laval, Quebec
  - Innovaderm Research, Montreal, Quebec
  - Centre de recherche dermatologique du Québec Métropolitain, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Infliximab: Placebo at weeks 0, 2, 8 during the first intervention period and infliximab 5mg/kg at weeks 14, 16 and 20 during second intervention period.
Period: First Intervention - Day 0 - Week 14
Arm/Group | Placebo Then Infliximab | Infliximab
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention Week 14 - Week 26
Arm/Group | Placebo Then Infliximab | Infliximab
Started | 12 (Patient withdrew at Week 14 and therefore never received infliximab.) | 12
Completed | 11 | 10
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Infliximab | Infliximab | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 1 | 3 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 49.92 (14.74) | 57.83 (12.42) | 53.87 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 12 | 24
Modified Palmoplantar Pustulosis Area and Severity Index (m-PPPASI) [Mean (Standard Deviation); unit: Units on a scale] — m-PPPASI = (E + I + D) Area X 0.2 (R palm) + (E + I + D) Area X 0.2 (L palm) + (E + I + D) Area X 0.3 (R sole) + (E + I + D) Area X 0.3 (L sole).
  Erythema, induration and desquamation are evaluated on a scale of 0 to 4 while area is evaluated on a scale of 0 to 6. The PPASI score can vary from 0 (absence of disease) to 72 (most severe palmoplantar psoriasis possible).
  Units on a scale | 26.7 (12.4) | 24.1 (11.4) | 25.4 (11.7)
Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: Units on a scale] — Impact on quality of life with the Dermatology Life Quality Index (DLQI) The aim of the questionnaire is to measure how much a patient's skin problem has affected their life over the previous week.
  * 0-1 = no effect at all on patient's life
  * 2-5 = small effect on patient's life
  * 6-10 = moderate effect on patient's life
  * 11-20 = very large effect on patient's life
  * 21-30 = extremely large effect on patient's life
  Units on a scale | 11.9 (6.9) | 9.8 (4.4) | 10.8 (5.8)
Physician's Global Assessment (PGA) [Mean (Standard Deviation); unit: Units on as scale] — Efficacy by comparing the mean Physician's Global Assessment(PGA).
  * 0 = clear
  * 1 = almost clear
  * 2 = Mild
  * 3 = Moderate
  * 4 = Severe
  * 5 = Very severe
  Units on as scale | 3.8 (0.6) | 3.5 (0.7) | 3.7 (0.6)
Palmoplantar Psoriasis Surface Area PPSA [Mean (Standard Deviation); unit: Percentage of affected area] — Efficacy by comparing the mean percent PPSA. The surface affected by psoriasis on palms and soles is estimated on the day of the visit as a percentage of the total surface of palms and soles affected by psoriasis. Each palm represents 20% and each sole 30%. As a rule of thumb half a palm equals 10% of the total surface area of palm and soles. A sole completely covered with psoriasis would have a PPSA of 30% (if the other sole and the palms are unaffected) while a palm completely covered with psoriasis would have a PPSA of 20% (if the other palm and the soles are unaffected).
  Percentage of affected area | 40.4 (21.6) | 37.1 (21.0) | 38.8 (20.9)

OUTCOME MEASURES:

1. Primary Outcome: 75% Improvement in Modified Palmoplantar Pustulosis Area and Severity Index (m-PPPASI) From Day 0
Description: Efficacy by comparing the number of patients reaching a 75% improvement in m-PPPASI (m-PPPASI 75) m-PPPASI = (E + I + D)Area X 0.2 (R palm) + (E + I + D) Area X 0.2 (L palm) + (E + I + D) Area X 0.3 (R sole) + (E + I + D) Area X 0.3 (L sole).
  Erythema, induration and desquamation are evaluated on a scale of 0 to 4 while area is evaluated on a scale of 0 to 6. The m-PPPASI score can vary from 0 (absence of disease) to 72 (most severe palmoplantar psoriasis possible).
Time Frame: 14 weeks
Population: The analysis was performed on the intent to treat (ITT) population. Nonresponder imputation (NRI) was used for patients who withdrew before the end of the study. They were treated as nonresponders from the point of withdrawal onward.
Measure: Number; unit: Participants
Arm/Group | Placebo Then Infliximab | Infliximab
Number analyzed (Participants) | 12 | 12
Participants | 1 | 4

2. Secondary Outcome: Number of Adverse Events at Week 14
Description: Safety of infliximab administered for 14 weeks in patients who received by comparing adverse events
Time Frame: 14 weeks
Measure: Number; unit: Adverse Events
Arm/Group | Placebo Then Infliximab | Infliximab
Number analyzed (Participants) | 12 | 12
Adverse Events | 20 | 32

3. Secondary Outcome: Mean Dermatology Life Quality Index (DLQI) at Week 14
Description: Impact on quality of life with the Dermatology Life Quality Index (DLQI) The aim of the questionnaire is to measure how much a patient's skin problem has affected their life over the previous week.
  * 0-1 = no effect at all on patient's life
  * 2-5 = small effect on patient's life
  * 6-10 = moderate effect on patient's life
  * 11-20 = very large effect on patient's life
  * 21-30 = extremely large effect on patient's life
Time Frame: 14 weeks
Population: The analysis was performed on the intent to treat (ITT) population and the imputation technique was last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Then Infliximab | Infliximab
Number analyzed (Participants) | 12 | 12
Units on a scale | 9.25 (7.23) | 4.50 (5.98)

4. Secondary Outcome: Mean Percent Palmoplantar Psoriasis Surface Area (PPSA) at Week 14
Description: Efficacy by comparing the mean percent PPSA. The surface affected by psoriasis on palms and soles is estimated on the day of the visit as a percentage of the total surface of palms and soles affected by psoriasis. Each palm represents 20% and each sole 30%. As a rule of thumb half a palm equals 10% of the total surface area of palm and soles. A sole completely covered with psoriasis would have a PPSA of 30% (if the other sole and the palms are unaffected) while a palm completely covered with psoriasis would have a PPSA of 20% (if the other palm and the soles are unaffected).
Time Frame: 14 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of affected area
Arm/Group | Placebo Then Infliximab | Infliximab
Number analyzed (Participants) | 12 | 12
Percentage of affected area | 38.58 (20.6) | 17.23 (15.75)

5. Secondary Outcome: Mean Physician's Global Assessment (PGA) at Week 14
Description: Efficacy by comparing the mean Physician's Global Assessment(PGA).
  * 0 = clear.
  * 1 = almost clear.
  * 2 = Mild.
  * 3 = Moderate.
  * 4 = Severe.
  * 5 = Very severe.
Time Frame: 14 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Then Infliximab | Infliximab
Number analyzed (Participants) | 12 | 12
Units on a scale | 3.33 (1.37) | 2 (0.95)

6. Secondary Outcome: Mean Percent Improvement in Modified Palmoplantar Pustulosis Area and Severity Index (m-PPPASI) at Week 26
Description: Efficacy of infliximab administered for 22 weeks in patients who received infliximab at Day 0 by evaluating the improvement over time in modified m-PPPASI from Day 0 to Week 26.
  m-PPPASI = (E + I + D)Area X 0.2 (R palm) + (E + I + D) Area X 0.2 (L palm) + (E + I + D) Area X 0.3 (R sole) + (E + I + D) Area X 0.3 (L sole).
  Erythema, induration and desquamation are evaluated on a scale of 0 to 4 while area is evaluated on a scale of 0 to 6. The m-PPPASI score can vary from 0 (absence of disease) to 72 (most severe palmoplantar psoriasis possible).
Time Frame: Baseline, 26 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent improvement
Arm/Group | Infliximab
Number analyzed (Participants) | 12
Percent improvement | 71.81 (31.59)

7. Secondary Outcome: Mean Percent Improvement in Dermatology Life Quality Index (DLQI) at Week 26
Description: Efficacy of infliximab administered for 22 weeks in patients who received infliximab at Day 0 by evaluating the improvement over time in dermatology life quality index (DLQI) from Day 0 to Week 26.
  Impact on quality of life with the DLQI. The aim of the questionnaire is to measure how much a patient's skin problem has affected their life over the previous week.
  * 0-1 = no effect at all on patient's life
  * 2-5 = small effect on patient's life
  * 6-10 = moderate effect on patient's life
  * 11-20 = very large effect on patient's life
  * 21-30 = extremely large effect on patient's life
Time Frame: Baseline, 26 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent improvement
Arm/Group | Infliximab
Number analyzed (Participants) | 12
Percent improvement | 63.45 (30.29)

8. Secondary Outcome: Mean Percent Improvement in Physician's Global Assessment (PGA) at Week 26
Description: Efficacy of infliximab administered for 22 weeks in patients who received infliximab at Day 0 by evaluating the improvement over time in Physician's Global Assessment (PGA) from Day 0 to Week 26.
  * 0 = clear
  * 1 = almost clear
  * 2 = Mild
  * 3 = Moderate
  * 4 = Severe
  * 5 = Very severe
Time Frame: Baseline, 26 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent improvement
Arm/Group | Infliximab
Number analyzed (Participants) | 12
Percent improvement | 47.92 (41.76)

9. Secondary Outcome: Mean Percent Improvement in Palmoplantar Psoriasis Surface Area (PPSA) at Week 26
Description: Efficacy of infliximab administered for 22 weeks in patients who received infliximab at Day 0 by evaluating the improvement over time in percent PPSA from Day 0 to Week 26. The surface affected by psoriasis on palms and soles is estimated on the day of the visit as a percentage of the total surface of palms and soles affected by psoriasis. Each palm represents 20% and each sole 30%. As a rule of thumb half a palm equals 10% of the total surface area of palm and soles.
Time Frame: Baseline, 26 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent improvement
Arm/Group | Infliximab
Number analyzed (Participants) | 12
Percent improvement | 65.91 (38.91)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all patients after the informed consent form was signed until the end of the study at week 26.
Description: Patients randomized to placebo then infliximab did not receive infliximab prior to week 14.
Groups:
- Infliximab: Infliximab 5mg/kg at weeks 0, 2, 6, 14 and 22 throughout the entire study.
Arm/Group | Infliximab | Placebo Then Infliximab
Serious Adverse Events (participants affected / at risk) | 2/12 | 1/12
Other Adverse Events (participants affected / at risk) | 11/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=12) | Placebo Then Infliximab (N=12)
Cellulitis Right Cheek (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sternum Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Caused by car accident
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=12) | Placebo Then Infliximab (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2)
Burn right arm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burning sensation to feet (Nervous system disorders) | 1 (3) | 0 (0)
Cellulitis Right Elbow (Infections and infestations) | 1 (1) | 0 (0)
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Common cold (Infections and infestations) | 3 (3) | 3 (4)
Costal ribs fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Erythema right forearm and both thighs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Facial flushing (Vascular disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 2 (3) | 1 (1)
Feet Oedema (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Ganglion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hair Loss (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Inflammed Seborrheic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Joint pain in hand (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Lower legs pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal reflux with pyrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain following dental surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Pain in foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain left shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pruritus right forearm and both thighs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Swelling left arm (General disorders) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vagal reaction (Nervous system disorders) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting and Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Worsening of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Worsening of hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The lack of validated scales to specifically assess severity of palmoplantar psoriasis. The study was powered to detect a difference of 55 percentage points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less